CLINICAL TRIAL: NCT01408264
Title: A Prospective Randomised Trial of 0.025 Wire Guided Cannulation Versus Current Practice 0.035 Wire Guided Cannulation
Brief Title: A Trial of 0.025 Wire Guided Cannulation Versus Current Practice 0.035 Wire Guided Cannulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WGC
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Abdominal Pain; Post-ERCP Acute Pancreatitis
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.035 guidewire (Active Comparator): conventional 0.035 guidewire
  Interventions: Device: Conventional 0.035 guidewire
- Olympus Visiglide 0.025 guidewire (Active Comparator): Olympus Visiglide 0.025
  Interventions: Device: Olympus Visiglide 0.025 guidewire

INTERVENTIONS:
Device: Conventional 0.035 guidewire — 0.035 guidewire
  Arms: 0.035 guidewire
Device: Olympus Visiglide 0.025 guidewire — 0.025 guidewire
  Arms: Olympus Visiglide 0.025 guidewire

SUMMARY:
The aim of this study is to determine whether using a smaller wire results in a higher success rate at endoscopic retrograde cholangiopancreatography (ERCP), and lower incidence of adverse events

DETAILED DESCRIPTION:
Cannulation of the bile duct is a prerequisite to successful therapeutic biliary endoscopy. Cannulation itself can carry substantial risk to the patient. Acute pancreatitis following ERCP can occur up to 5% of cases. The risk increases in patients with non dilated bile ducts, young age, known past history of pancreatitis and suspected sphincter of oddi dysfunction. During the procedure of ERCP, the number of pancreatograms also correlates with incidence of post ERCP pancreatitis. Hydrostatic pressure by contrast injection into the pancreatic duct may be the principal cause of pancreatitis. We performed a meta-analysis of randomized controlled trials that compared the technique of contrast guided to wire guide cannulation in achieving bile duct cannulation during ERCP and found that wire guide cannulation was better at the prevention of post ERCP pancreatitis. The use of a guide wire obviates the need for contrast injection. The current standard is the use of a 0.035" guidewire with a hydrophilic tip. We now postulate that the use of a 0.025" further reduces post-ERCP pancreatitis as a finer wire theoretically induces less trauma to the pancreatic orifice.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for ERCP who have an intact naïve papilla are considered for inclusion

Exclusion Criteria:

* Age <18yrs
* Acute illness (hypotension: BP<90mmHg, hypoxia: O2 <95%, haemodynamic instability)
* Inability or refusal to give informed consent.
* Patients with previous sphincterotomy
* Pancreatic or ampullary cancer are excluded as post-ERCP pancreatitis (PEP) is very uncommon in these subgroups and tumour-related anatomical variation may alter cannulation technique.

(consider substratify results for this subgroup, but exclude if duodenal stenosis precludes an attempt on the papilla)

* Patients with surgically altered anatomy (Bilroth II gastrectomy and Roux en Y anastomosis) are excluded as cannulation technique is fundamentally different from that in normal anatomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | 30 days after ERCP
  Reported post-ERCP pancreatitis

SECONDARY OUTCOMES:
Abdominal pain | 30 days after ERCP
  Abdominal pain
Prolonged hospitalisation | 30 days after ERCP
  Prolonged hospitalisation
Death | 30 days after ERCP
  Death

CONTACTS AND LOCATIONS:
Overall Officials: James Y Lau, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Bassan MS, Sundaralingam P, Fanning SB, Lau J, Menon J, Ong E, Rerknimitr R, Seo DW, Teo EK, Wang HP, Reddy DN, Goh KL, Bourke MJ. The impact of wire caliber on ERCP outcomes: a multicenter randomized controlled trial of 0.025-inch and 0.035-inch guidewires. Gastrointest Endosc. 2018 Jun;87(6):1454-1460. doi: 10.1016/j.gie.2017.11.037. Epub 2018 Jan 6. PMID 29317269